CLINICAL TRIAL: NCT00846300
Title: An Intervention to Improve Medication Knowledge & Compliance Among Family Practice Patients in South Texas: An RRNEST Study.
Brief Title: A Brief Intervention to Improve Medication Knowledge and Adherence Among Family Medicine Patients in South Texas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sandra Burge, Ph.D., UTHSCSA
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HP000016-01
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus, Type 2; Hyperlipidemia; Hypertension
Keywords: Patient compliance; Hispanics; Health Behavior; Family Physicians; Primary Healthcare
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperlipidemias; Hypertension; Patient Compliance; Health Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Physician counseling for health behavior change — Physician counseling for health behavior change, compared to a no-counseling comparison group

SUMMARY:
This study examines a brief physician counseling intervention to improved medication knowledge and compliance in family medicine patients who have diabetes, hypertension or high cholesterol.

DETAILED DESCRIPTION:
This study examined a brief intervention to improve medication knowledge and compliance in family medicine patients. The study was conducted in a network of six family medicine residency programs in South Texas, funded by a grant from the Health Research Services Administration. Family medicine patients were invited to participate in the study if they took medicines for type 2 diabetes, hypertension, or hyperlipidemia and responded "yes" to the screening question: "Do you sometimes have trouble taking all your medications as prescribed?"

At enrollment, clinic staff administered a Medication Survey to patients to assess the variables: readiness to change, reported medication knowledge; reported compliance, and predictors of knowledge and compliance. Self-reports of compliance were validated with a social desirability scale, and with physician impressions. Six and twelve weeks post-enrollment, interviewers administered followup surveys by telephone to assess change over time in medication knowledge and compliance. One year post-enrollment, investigators conducted a chart review to examine changes in health outcomes: blood pressure or HbA1c or cholesterol levels, and number of hospitalizations.

Three physicians per clinic site (18 total) conducted medication interventions for the purpose of this study. This intervention was brief behavior change counseling done in the context of a routine office visit, guided by simple strategies outlined in Rollnick et al (1999). First, physicians reviewed subjects= medication regimen and addressed their concerns. We selected a simple strategy from Rollnick et al. - a brainstorming session - that built patients' confidence to change health behaviors. Afterward, physicians offered pillboxes to patients who desired them, and reviewed potential adverse reactions to medicines. One week after the intervention, physicians telephoned patients to reinforce behavior change and to answer questions about the medications. Prior to training physicians to conduct this intervention, we enrolled five subjects per physician into a control group. We attempted to blind physicians to these patients= enrollment status; usual care was provided to control subjects. After training, enrollees' charts were flagged so that physicians knew to conduct the intervention. We sought five patients per physician to receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sometimes has trouble taking medicines as they're prescribed
* Has diabetes type 2, or hypertension, or high cholesterol for which they take prescription medicines
* Is a patient of 18 doctors conducting the intervention

Exclusion Criteria:

* Subjects under age 18

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2001-08; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Change in self-reported medication knowledge | 6 and 12 weeks post-intervention
Change in self-reported medication compliance | 6 and 12 weeks post intervention
Change in HbA1c for patients with Diabetes | 1 year post intervention
Change in Lipids | 1 year post intervention
Change in blood pressure | 1 year post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Burge, Ph.D., Principal Investigator — University of Texas Health Science Center San Antonio
Locations (6):
- United States (6):
  - Christus Memorial Hospital, Corpus Christi, Texas
  - Valley Baptist Family Medicine Residency Program, Harlingen, Texas
  - Laredo Medical Group, Laredo, Texas
  - McAllen Family Medicine Residency Program, McAllen, Texas
  - Family Medicine Residency Program, Christus Santa Rosa Hospital, San Antonio, Texas
  - Dept Family & Community Medicine, UTHSCSA, San Antonio, Texas